CLINICAL TRIAL: NCT06417801
Title: PANGEIA-2: Prevalence of Emerging Treatment-induced Mutations in metastaticER Positive Breast Cancer.
Brief Title: Prevalence of Emerging Treatment-induced Mutations in Metastatic ER-positive Breast Cancer.
Acronym: Pangeia-2
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D3612L00003
Record Dates: First submitted 2024-05-13; First posted 2024-05-16 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Breast Cancer
Keywords: Breast Cancer; ER-positive; ESR-1 mutation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue.

GROUPS / COHORTS (2):
- Cohort 1 (N=30): Locally-advanced/metastatic HR+/HER2- breast cancer, either treatment naive or previously exposed to adjuvant therapies, no prior palliative therapy, candidates to receive first-line hormone therapy, primary tumor tissue available.
- Cohot 2 (N=40): Locally-advanced/metastatic HR+/HER2- breast cancer, progression during hormone therapy plus CDK inhibitor; primary tumor tissue available.

SUMMARY:
Observational study on prevalence of emerging ESR1 mutations in liquid biopsy in two cohorts of patients with breast cancer (with and without prior therapies in metastatic setting) in comparison with patient's baseline ESR1 mutation status as defined by tissue profiling.

DETAILED DESCRIPTION:
This is a prospective observational biomarker cohort study. Biomarkers: GS Focus Liquid Breast (liquid biopsy sequencing assay, covers mutations in ESR1, PIK3CA, AKT1, PTEN, ERBB2, BRCA1, BRCA2, PALB2) and parallel GS Focus Breast (tissue sequencing assay performed in baseline tissue biopsy from primary tumor or metastatic lesion not exposed to any systemic therapy, cover same gene panel).

Biomarker assessment will be carried out by NGS methodology in both liquid biopsy and baseline tissue biopsy. Both strategies consider a custom panel covering PIK3CA, AKT1, PTEN, ESR1, BRCA1, BRCA2, PALB2, ERBB2 genes.

NGS panels were internally validated and presented sensitivity, specificity and accuracy of 100,00% with a limit of detection of 0,5% VAF for liquid biopsy panel and sensitivity, specificity and accuracy of 100,00% with a limit of detection of 5% VAF for tissue panel. Basically, DNA is extracted from tissue samples (FFPE) and plasma using QIASymphony extractions kits. An input of 10 and 100 ng is required for liquid biopsy and tissue respectively. NGS libraries is prepared using QIAseq Targeted DNA Custom Panel (QIAGEN). Sequencing is performed in Illumina platform (NextSeq for liquid biopsy and MiSeq for tissue samples) in paired-end 2x 150 cycles.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1:

* BC patients, male and female, 18 years old and older, pre or post menopausal, with HR+ (ER and/or PR positive), Her-2 negative (confirmed centrally) locally advanced irresectable and/or metastatic disease
* Confirmation of HR and Her-2 status may be performed in the primary tumor or in the metastatic lesion (patients with discordant results may be included)
* Patients must be candidates to CDK4/6i therapy in combination with endocrine therapy in the first line setting (with or without ovarian suppression)
* Patients may have received one previous line of chemotherapy in the metastatic setting, but no endocrine therapy in the metastatic setting is allowed
* Patients may have received chemotherapy in the neo/adjuvant setting
* Patients may have received endocrine therapy (with or without ovarian suppression) in the neo/adjuvant setting
* Patients may have received a CDK4/6i in the adjuvant setting, provided they are still candidates for CDK4/6i therapy in the metastatic setting
* Patients must be able to undergo a liquid biopsy procedure before starting their first line treatment
* All patients must fill and sign an informed consent form.

Cohort 2:

* BC patients, male and felame, 18 years old and older, pre or post menopausal, with HR+ (ER and/or PR positive), Her-2 negative (confirmed centrally) locally advanced irresectable and/or metastatic disease who have progressed on a CDK4/6i in combination with endocrine therapy (with or without ovarian suppression) in the first or second line setting
* All other non-conflicting inclusion criteria for cohort 1 apply.

Exclusion Criteria:

Patients with HR+ (ER and/or PR positive) and Her-2 negative disease NOT confirmed centrally

* Patients with NO radiologic and/or pathologic confirmed locally irresectable and/or metastatic breast cancer
* Patients who are NOT candidates for further systemic treatment after diagnosis of metastatic disease or disease progression
* Patients who have already started a CDK4/6i in combination with endocrine therapy (with or without ovarian suppression) for metastatic disease in the first line setting (for cohort 1); and patients who have already started a new line of treatment for metastatic disease after disease progression on a CDK4/6i in combination with endocrine therapy (with or without ovarian suppression)(for cohort 2)
* Patients who are NOT able to undergo a liquid biopsy procedure
* Patients who are NOT able to provide informed consent.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Two parallel cohorts:
  1. locally-advanced/metastatic HR+/HER2- breast cancer, either treatment naive or previously exposed to adjuvant therapies, no prior palliative therapy, candidates to receive first-line hormone therapy, primary tumor tissue available;
  2. locally-advanced/metastatic HR+/HER2- breast cancer, progression during hormone therapy plus CDK inhibitor; primary tumor tissue available.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-06-17 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of emerging ESR1 mutations | Aug, 2024
  To define the prevalence of emerging ESR1 mutations in liquid biopsy in two cohorts of BC patients (with and without prior therapies in metastatic setting) and compare with patient's baseline ESR1 mutation status as defined by tissue profiling.

SECONDARY OUTCOMES:
Define the prevalence of PIK3CA, AKT1, PTEN, BRCA1, BRCA2, PALB2, ERBB2 mutations. | Aug, 2024
  To define the prevalence of PIK3CA, AKT1, PTEN, BRCA1, BRCA2, PALB2, ERBB2 mutations in liquid biopsy and compare with patient's baseline status.

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Dienstmann, Principal Investigator — Oncoclínicas
Locations (1):
- Research Site, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/